CLINICAL TRIAL: NCT03231410
Title: Role of Monocytes Adhesion and Vascular Lesions in Vascular Access Success or Failure in Uremic Patients
Acronym: ROMAVAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wroclaw Medical University (Other)
Collaborators: Universitätsklinikum Halle (Unknown)
Responsible Party: Principal Investigator, Tomasz Gołębiowski, MD, PhD, Wroclaw Medical University
Other Study IDs: WroclawMU
Record Dates: First submitted 2017-07-16; First posted 2017-07-27 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: End Stage Renal Disease; Arteriovenous Fistula
Keywords: arteriovenous fistula; maturation; monocyte adhesion; vascular access
MeSH Terms: conditions — Kidney Failure, Chronic; Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Transcripts of genes related to calcification (osteopontin, osteokalcin, RunX2), inflammation (TNFa, IL6) and atherosclerosis (ACE/ACE2, VCAM-1, ICAM-1) processes will be assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is designed to identify novel predictors of vascular access success or failure in chronic kidney disease patients. Despite efforts to improve placement of arteriovenous fistula (AVF) the primary failure rates are reported as high as 20-50%, but standard tools like ultrasound cannot inform the clinician sufficiently to accurately predict success or failure.

The aim of this study is to perform enhanced assessments of arterial health preoperatively and correlate these measurements with vascular lesions (microscopic tissue changes and monocyte infiltration) and early AVF outcome.

Activation of monocytes in uremia condition is responsible for endothelium dysfunction, intimal hyperplasia and atherosclerosis. The investigators expect that stiff arteries caused by monocyte dysfunction refer to the poor distensability and probably longer maturation time.

DETAILED DESCRIPTION:
Research Project Objectives

For patients with progressive chronic kidney disease the definitive treatment is a renal replacement therapy. One of the methods is hemodialysis, which is frequently chosen in patients above 65y. of age. Several clinical practice guidelines recommend an arteriovenous fistula (AVF), rather than a central venous catheter or arteriovenous graft, as the preferred access for maintenance hemodialysis (HD) therapy. Despite efforts to improve placement of AVF in both the hemodialysis incident and prevalent population, many patients continue dialysis through a central venous catheter, exposing them to higher risks of infection, co-morbidity and mortality in comparison to use an AVF for HD. Furthermore, AVF primary failure rates are reportedly as high in 20-50% in published series confirming that ultrasound cannot sufficiently inform the clinician to accurately predict success or failure. Because of higher risk of early AVF failure offering this type of access is questionable in diabetics, unfavorable artery/vein diameter and elderly people. To perform hemodialysis vascular access ensuring adequate blood flow is required. Such access is most commonly obtained by the creation of the vascular connection between an artery and a vein on the upper limb. Recent data from European and National registries clearly indicate huge increase of incident dialysis patients above 65y. In older patients with many co-morbidities and limited predictive survival decision whether to start dialysis, when and how should be cautious. When choosing vascular access fistula non-maturation problem must be taken into account. The successful creation of a permanent vascular access depends on vessel health, patient characteristics and possibly genetic factors. In patients with end stage renal disease circulating monocytes are activated and proinflammatory monocytes are expanded. Recent data indicates that uremic conditions drive monocytes to differentiate and interact with artery wall promoting atherosclerosis. This interaction can be studied in the laboratory by testing inﬂammatory activity of THP-1 monocytes and by checking proatherosclerotic and calcification markers in the artery specimen (taken during AVF creation).

Research hypothesis: monocytes activation and advancement of vascular lesions affect the process of remodeling (maturation) of arteriovenous fistula, determines its usability (functionality). The investigators also hypothesize that an increase in the collagen content of the vascular media (medial fibrosis) preoperatively would impair vascular dilation and thereby, limit the postoperative increase in arteriovenous fistula diameter, blood flow and finally AVF maturation.

Working second hypothesis: the metrical age of patient with mild to moderate vascular lesions is not limiting factor in AVF success rate and maturation.

The main aim of the study is assessment of changes in the vessels and monocyte activation and its impact on the ability to create AVF and its usability for hemodialysis. Secondary objective of this study is to perform enhanced assessments of arterial health preoperatively and correlate these measurements with vascular lesions. The investigators intend to perform preoperative vascular mapping, flow mediated dilatation (FMD) and assess endothelial function. These non invasive measurements will provide a more accurate picture of overall vascular health prior to AVF formation with the ultimate intention of informing the clinician as to the likelihood of success or failure.

Work plan

Participants will be subjects of a thorough evaluation of the morphological and functional state of upper limb vessels by the techniques presented in the methodology of the study. The study plan foresees the recruitment of patients, whose will have their vessels of the upper limbs carried out in-depth assessment. Then creation of the vascular access - arteriovenous fistula for dialysis, will be performed. Arterial and venous specimens will be sampled during arteriovenous fistula surgery. Its maturation will be evaluated in a conventional manner (functional fistula allowing delivery of adequate dialysis dose) as well as using criteria mentioned in the publications.

Study design Prospective study with recruitment of consecutive approximately 30 patients with chronic kidney disease stage 4 or 5, who will be referred for vascular access creation for hemodialysis.

Inclusion: (1) Aged >18 years, (2) Has chronic kidney disease with estimated glomerular filtration rate (eGFR) <20 mL/min/1.73 m2 , (3) Is undergoing AVF creation with venous end-to-arterial side anastomosis in the upper extremity.

Exclusion: (1) Heart failure of New York Heart Association functional class III or IV, and (2) Episode of cardio- or cerebrovascular event or receiving intervention therapy within 3 months prior to screening. The need for any interventional procedure (surgery or angioplasty) to correct an occlusive or malfunctioning fistula.

After obtaining an informed consent to participate in the study each participant will be tested with followed measures.

Study measures

Demographic and clinical characteristic will be collected during interview (family longevity, hospitalizations, history of vein cannulation) and based on medical records (cardiac events including angiographic studies, cancer, diabetes, peripheral artery diseases, dementia and other co-morbidities. Physical examination focused on heart function (blood pressure in two positions, heart rate, congestion in auscultation and chest as well as vascular anatomy examination with Allen test (patency of palmar arch), pulse presence, veins patency with and without stasis.

Imaging studies

Ultrasound condition of vessel will be evaluated prior AVF creation (upper arms flow, diameter of arteries and veins, possible stenosis, etc) and in follow up period (day 1, 14, 30). In selected cases (history of previous subclavian vein catheterization, collateral circulation developed) venography will be performed.

Histomorphology and immunomorphology of the vessels

Arterial and venous specimens will be stained. Following markers will be used for immunomorphology assessment. Pro-atherosclerotic molecules (ACE/ACE2, VCAM-1, ICAM-1) expression in artery and vein (1-2mm section taken during surgery) which undergo immediate freezing. Masson's trichrome-staining of samples will be used to quantify medial fibrosis (collagen) both the artery and the vein.

Whole blood parameters for circulating molecules/cells

Blood samples will be taken at routine control, or before routine dialysis session in HD patients (referred for AVF placement). Samples will be collected and stored before the AVF. Following vascular biomarkers will be assessed by enzyme-linked immunosorbent assays:ADMA and sICAM1, sVCAM1. For HO-1 gene polymorphism genotyping blood sample will be collected ones. It will be evaluated by Real Time PCR (frozen DNA samples).

Leukocytic RNA, serum and isolation of primary human monocytes

Blood samples for RNA and serum isolation will be obtained from ESRD/HD patients. Blood samples for leukocytic RNA isolation will be drawn into Tempus Blood RNA Tubes (Life Technologies). Total RNA is isolated with Tempus Spin RNA Isolation Kits according to the manufacturer's instructions (Life Technologies). Transcripts of genes related to calcification (osteopontin, osteokalcin, RunX2), inflammation (TNFa, IL6) and atherosclerosis (ACE/ACE2, VCAM-1, ICAM-1) processes will be assessed.

Adhesion and transmigration assays

Another in vitro test is designed for adhesion/invasion of THP-1 monocytes. It will test aggressive properties of monocytes infiltration endothelium. Adhesion of THP-1 monocytes to endothelial HUVEC monolayers and all transmigration assays will be performed.

Vascular Functional tests

A number of measures are available to assess vascular function (and predict cardiovascular risk) such as flow mediated dilation (FMD) or peak blood flow (PBF) of the brachial artery. FMD provides an assessment of macrovascular endothelial cell function. Healthy endothelium releases a potent vasodilator (nitric oxide, NO) in response to ischemic stress such as cuff occlusion of the brachial artery. FMD is a measure of the change in the brachial artery diameter in response to cuff occlusion and subsequent NO release. Whereas FMD reflects the ability of a large artery to vasodilate, the subsequent change in blood flow that ensues represents the health of the peripheral resistance vessels or microvascular function.

Above mentioned vascular tests will be conducted to assess endothelial dysfunction. The absolute increase in diameter after ischemia (BAD, brachial artery diameter), peak blood flow (PBF) and flow-mediated dilation (FMD) will be performed on both arms at day 0 (pre AVF creation), and then at day 1, 14-28 (opposite to AVF arm). The measurement will be performed according to published standard protocol for FMD measurement using Aloka alpha 7 USG device with Doppler linear probe.

Routine laboratory parameters collected at baseline and during follow-up (14-28, 56-60, 90 day): Complete blood counts with focus on neutrophil-lymphocyte ratio (NLR), phosphorus, calcium, PTH, C-reactive protein (CRP), urea acid, lipids (cholesterol fractions, triglycerides).

Statistical analysis

All participants data from recruitment and follow up will be collected in special designed computer program. The primary outcome of this study is AVF success (patent and mature) at 8 and 14 weeks post creation. Baseline patient characteristics including age, gender and co-morbidities will be compared between the patients with successful AVF and those with unsuccessful AVF. Categorical variables will be presented by frequency (percentage) and comparisons will be made via the Chi-square or Fisher's Exact test. Underlying distributions of continuous variables will be tested for normality using the Shapiro-Wilk test and then analyzed with appropriate tests. All analyses will be performed by external statistical laboratory with high references. The professional statistical expertise is planned (PREST laboratory at Mathematical Institute in Wroclaw) with utilization of R package and STATISTICA 10 software.

ELIGIBILITY:
Inclusion Criteria:

* aged >18 years,
* chronic kidney disease with estimated glomerular filtration rate (eGFR) <20 mL/min/1.73 m2,
* undergoing AVF creation with venous end-to-arterial side anastomosis in the upper extremity.

Exclusion Criteria:

* Heart failure of New York Heart Association functional class III or IV,
* Episode of cardio- or cerebrovascular event or receiving intervention therapy within 3 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Prospective study with recruitment of consecutive 30 patients with chronic kidney disease stage 4 or 5, who will be referred for vascular access creation for hemodialysis.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Primary patency rate | Baseline to 12 months after AVF creation
  Primary patency rate

SECONDARY OUTCOMES:
Hemodialysis AVF blood flow | Baseline to 12 months after AVF creation
  Blood flow by Doppler ultrasound on brachial artery (ml/min.)

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Gołębiowski, MD, PhD, Principal Investigator — Department of Nephrology and Transplantation Medicine, Wroclaw Medical University; Mariusz Kusztal, MD, PhD, Study Director — Department of Nephrology and Transplantation Medicine, Wroclaw Medical University; Krzysztof Letachowicz, MD, PhD, Study Chair — Department of Nephrology and Transplantation Medicine, Wroclaw Medical University
Locations (1):
- Department of Nephrology and Transplantation Medicine, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tordoir J, Canaud B, Haage P, Konner K, Basci A, Fouque D, Kooman J, Martin-Malo A, Pedrini L, Pizzarelli F, Tattersall J, Vennegoor M, Wanner C, ter Wee P, Vanholder R. EBPG on Vascular Access. Nephrol Dial Transplant. 2007 May;22 Suppl 2:ii88-117. doi: 10.1093/ndt/gfm021. No abstract available. PMID 17507428
- [Background] Roy-Chaudhury P, Kelly BS, Melhem M, Zhang J, Li J, Desai P, Munda R, Heffelfinger SC. Vascular access in hemodialysis: issues, management, and emerging concepts. Cardiol Clin. 2005 Aug;23(3):249-73. doi: 10.1016/j.ccl.2005.04.004. PMID 16084276
- [Background] Trojanowicz B, Ulrich C, Seibert E, Fiedler R, Girndt M. Uremic conditions drive human monocytes to pro-atherogenic differentiation via an angiotensin-dependent mechanism. PLoS One. 2014 Jul 8;9(7):e102137. doi: 10.1371/journal.pone.0102137. eCollection 2014. PMID 25003524
- [Background] Himmelfarb J. Uremic toxicity, oxidative stress, and hemodialysis as renal replacement therapy. Semin Dial. 2009 Nov-Dec;22(6):636-43. doi: 10.1111/j.1525-139X.2009.00659.x. PMID 20017834
- [Background] Zickler D, Willy K, Girndt M, Fiedler R, Martus P, Storr M, Schindler R. High cut-off dialysis in chronic haemodialysis patients reduces serum procalcific activity. Nephrol Dial Transplant. 2016 Oct;31(10):1706-12. doi: 10.1093/ndt/gfw293. Epub 2016 Jul 20. PMID 27445317
- [Background] Stoner L, Sabatier MJ. Use of ultrasound for non-invasive assessment of flow-mediated dilation. J Atheroscler Thromb. 2012;19(5):407-21. doi: 10.5551/jat.11395. Epub 2012 Mar 1. PMID 22659525
- [Background] Yilmaz MI, Stenvinkel P, Sonmez A, Saglam M, Yaman H, Kilic S, Eyileten T, Caglar K, Oguz Y, Vural A, Cakar M, Altun B, Yenicesu M, Carrero JJ. Vascular health, systemic inflammation and progressive reduction in kidney function; clinical determinants and impact on cardiovascular outcomes. Nephrol Dial Transplant. 2011 Nov;26(11):3537-43. doi: 10.1093/ndt/gfr081. Epub 2011 Mar 4. PMID 21378154